CLINICAL TRIAL: NCT01782924
Title: An Extension Study in Subjects With Plaque Psoriasis
Brief Title: A Phase 3 Clinical Study of KHK4827
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 4827-003
Record Dates: First submitted 2013-01-27; First posted 2013-02-04 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — brodalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK4827 140mg SC (Experimental)
  Interventions: Drug: KHK4827
- KHK4827 210mg SC (Experimental)
  Interventions: Drug: KHK4827

INTERVENTIONS:
Drug: KHK4827

SUMMARY:
This study is designed to evaluate safety and efficacy of long-term exposure of KHK4827 in subjects with moderate to severe plaque psoriasis who have completed the preceding Study 4827-002.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed the written informed consent form to participate in this study
* Subject has completed the week 12 evaluation of Study 4827-002

Exclusion Criteria:

* Subject has had a serious infection, defined as requiring systemic treatment with antibiotics or antivirals (excluding oral administration)
* Subject has been judged to be ineligible for participation in the study by the investigators/subinvestigators

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence and types of adverse events and adverse reactions | 52 weeks
Laboratory values and vital signs | 52 weeks
Development of anti-KHK4827 antibody | 52 weeks

SECONDARY OUTCOMES:
Percent improvement from baseline in Psoriasis Area and Severity Index (PASI) | 52 weeks
A 50% improvement in PASI (PASI 50), PASI 75, PASI 90 and PASI 100 response | 52 weeks
Static physician's global assessment (sPGA) of "clear or almost clear (0 or 1)" | 52 weeks
sPGA of "clear (0)" | 52 weeks
Body surface area involvement (BSA) of lesion | 52 weeks
American College of Rheumatology (ACR) 20 (only in subjects with psoriasis arthritis) | 52 weeks
Profiles of pharmacokinetics | 52 weeks
  Concentration of KHK4827 in serum

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Chiyoda-ku, Tokyo, Japan